CLINICAL TRIAL: NCT04985188
Title: Quantitative Ultrasound Imaging Parameters for Hepatic Steatosis in Patients With Non-alcoholic Fatty Liver Disease: Multicenter Prospective Study
Brief Title: Quantitative Ultrasound for Diagnosing Hepatic Steatosis in Nonalcoholic Fatty Liver Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Ruijin Hospital (Other); Shenzhen Second People's Hospital (Other); Samsung Medison (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: 2102-159-1199
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative ultrasound (QUS) technique — Measurement of quantitative ultrasound parameter using clinical US machine (RS85)

SUMMARY:
To evaluate the diagnostic performance of quantitative ultrasound parameters for assessing hepatic steatosis in non-alcoholic fatty liver disease using histologic results as reference standard

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected or proven nonalcoholic fatty liver disease (NAFLD)
* Patients who are scheduled hepatic parenchymal biopsy for suspected liver disease or hepatectomy for living donor liver donation
* aged ≥ 18 years who are willing and able to complete all procedures

Exclusion Criteria:

* excessive alcohol consumption within 2 years (40g/day for men, 20g/day for women)
* clinical, laboratory, or histologic evidence of a liver disease other than NAFLD, including viral hepatitis, autoimmune hepatitis, or genetic or acquired disorders
* use of steatogenic or hepatotoxic medication
* evidence of decompensated liver disease
* history of liver surgery
* any other condition believed by investigator to affect a patients' compliance, or completion of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinically suspected or proven nonalcoholic fatty liver disease (NAFLD)
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-08-12 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of quantitative ultrasound parameters for diagnosing hepatic steatosis (S1) | 1 month
  Evaluation of area under the ROC curve (AUC) for the detection of fatty liver (S1)(reference standard: pathologic result)

SECONDARY OUTCOMES:
Diagnostic performance of quantitative ultrasound parameters for diagnosing hepatic steatosis (S2 and S3) | 1 month
  Evaluation of area under the ROC curve (AUC) for the detection of fatty liver (S2 and S3)(reference standard: pathologic result)
Diagnostic performance of quantitative ultrasound parameters for diagnosing nonalcoholic steatohepatitis (NASH) | 1 month
  Evaluation of area under the ROC curve (AUC) for the detection of nonalcoholic steatohepatitis (reference standard: pathologic result)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang TY, Li ZY, Tian J, Xie XJ, Lee JM, Ren XP, Xie XY. Metabolic Dysfunction-Associated Steatotic Liver Disease at Quantitative US: International Prospective Study. Radiology. 2025 Jul;316(1):e242564. doi: 10.1148/radiol.242564. PMID 40662970